CLINICAL TRIAL: NCT00224692
Title: MK III Trial: Analgesic Effect in Children of Low-Dose Ketamine for Mucositis Treated by Patient-Controlled Analgesia With Morphine
Brief Title: Analgesic Effect in Children of Low-Dose Ketamine for Mucositis Treated by Patient-Controlled Analgesia With Morphine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P010918; CRC01022
Record Dates: First submitted 2005-09-19; First posted 2005-09-23 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Cancer; Mucositis
Keywords: Mucositis; Pain; Morphine; Ketamine
MeSH Terms: conditions — Neoplasms; Mucositis; Pain | interventions — Ketamine

INTERVENTIONS:
Drug: Low dose ketamine

SUMMARY:
Hypothesis : Low dose ketamine has an analgesic effect in children with mucositis treated by patient-controlled analgesia with morphine

DETAILED DESCRIPTION:
Double blind versus placebo multicenter Phase III trial of kétamine in children with chemotherapy induced-mucositis treated by patient-controlled analgesia with morphine

ELIGIBILITY:
Inclusion Criteria:

* Painful mucositis
* Child from 5 to 18 years.
* Presenting mucitis induced by chemotherapy or a conditioning of graft hematopoïetic.
* A pain not controlled by systematic paracetamol (10mg/kg/4h) or a the propacetamol (20mg/kg/4h).
* Not presenting a neurological or psychological difficulty at the use of the PCA or a EVA.
* First morphine amount going back to less 48h, and lass administration dating of more than 4h at the time of the beginning of the perfusion of Ketamine/placebo (EVA > 30 after stop morphine).
* Assent signed by the parents and each time possible by the child.

Exclusion Criteria:

* The child was already included in the study.
* The age of psychomotor development is lower than 5 years
* Presence of a depression or a major depressive episode according to definition DSM IV.
* Hepatic or renal anomaly major (rank 3 or 4 of the scale of toxicity NCI CTC v2.0)
* Bilirubin>3N
* Gamma WP>3N
* SGOT or SGPT >5N
* Creatinin>3N

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2003-02; Study Completion 2006-08

PRIMARY OUTCOMES:
Pain score

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne JACQZ-AIGRAIN, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré Service Pédiatrie-Hémato-immunologie, Paris, Île-de-France Region, France